CLINICAL TRIAL: NCT04137458
Title: Exploration of the the Relationship Between Inflammation and Integrity of the Blood-brain Barrier in Suicidal Behaviour
Brief Title: Exploration of the Relationship Between Inflammation and Integrity of the Blood-Brain Barrier in Suicidal Behaviour
Acronym: IBIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL19_0227; 2019-A01277-50 (Other: ANSM)
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Depression
Keywords: Psychiatry; Blood Brain Barrie; Suicide attempt; Inflammation
MeSH Terms: conditions — Depression; Suicide, Attempted; Inflammation | interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): The investigator will withdraw biological samples and a biological and DNA bank will also be realized
  Interventions: Biological: Biological analysis

INTERVENTIONS:
Biological: Biological analysis — Blood and salivary samples will be taken at inclusion and a psychiatric assessment will be carried out

SUMMARY:
Recent studies have revealed an association between history of suicide attempt and inflammatory markers in both the cerebrospinal fluid and the plasma. Post mortem studies have shown an increase in microglial activation in the brain tissue of suicide victims. However the relationship between peripheral and central inflammation in suicide is probably mediated by complex biological processes that are yet elucidated. An increase of blood S100B levels (biomarker of neurovascular damage; PMID 14530574) has been reported in adolescents with suicidal ideation vs. controls and independently of psychiatric disorder. The investigators hypothesize that peripheral inflammation may alter BBB which normally acts as a filter to ensure proper neuronal functioning in suicidal vs. non suicidal patients.

DETAILED DESCRIPTION:
105 participants will be recruited :

* 35 depressed patients having attempted suicide (maximum 3 attempts in life)
* 35 depressed patients without history of suicide attempt (affective controls)
* 35 healhy controls with no lifetime psychiatric history.

Only one visit is planned. A clinical assessment (2 hours) will be performed to characterise pschopathology and suicidal characteristics. Blood and salivary samples will be obtained in order to measure inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* Able to understand nature, aims, and methodology of the study

Depending on the population :

* Current depressive episode (according to DSM-5 criteria) with a recent suicide attempt (within the 8 days before inclusion) and no more than 3 attempts in life
* Current depressive episode (according to DSM-5 criteria) without suicide attempt
* No psychiatric history (according to DSM-5 criteria)

Exclusion Criteria:

* Inflammatory diseases or intercurrent infections, or chronic diseases such as hepatitis C or B, HIV, Alzheimer's, cancer or autoimmune disease
* Current antibiotic or anti-inflammatory treatments
* Refusal to participate
* Lifetime Schizoaffective disorder or schizophrenia
* On protective measures (guardianship or trusteeship)
* Deprived of liberty subject (administrative decision)
* In exclusion period for another protocol
* Not affiliated to a social security agency
* Unable to understand and/or answer a questionnaire
* Pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Blood level of S100B | at inclusion
  Blood level of S100B measured in 3 groups (i.e. suicide attempters, affective controls, healthy controls)

SECONDARY OUTCOMES:
Determination of leukocyte signature associated with suicidal behavior and depression | at inclusion
  Comparison of the number and percentage of leukocytes (lymphocytes, monocytes, neutrophils) in the blood between the 3 patients groups
Profile of peripheral inflammation of each group | at inclusion
  Characterization of activation state of leukocytes of CD4 / CD8 (T cells), NK cells, CD14 / CD33 (monocytes / macrophages)
Identification of general peripheral inflammation | at inclusion
  Between groups comparison of blood levels of CRP
Pro-inflammatory profile based on cytokins of each group | at inclusion
  Serum pro-inflammatory interleukins (IL) -1b, IL2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-9, IL-10, IL-12, IL-13 , TGF-b, interferon IFN-g, TNF-a, TNF-b
Profile of salivary interleukins | at inclusion
  Profile of salivary interleukins Il-6, Il-13 et Il-17 within and between groups
Serum levels of glial fibrillary actin protein (GFAP) | at inclusion
  Between group comparison of serum levels (ng / ml) of glial fibrillary actin protein (GFAP)
Serum levels of specific neuronal enolase (NSE) | at inclusion
  Between group comparison of serum levels (ng / ml) of specific neuronal enolase (NSE)
Serum levels of ubiquitinar-carboxy-terminal hydrolase L1 (UCH-L1) | at inclusion
  Between group comparison of serum levels (ng / ml) of ubiquitinar-carboxy-terminal hydrolase L1 (UCH-L1)
Salivary levels of S100B protein | at inclusion
  Between group comparison of salivary levels of S100B protein
Salivary levels of specific neuronal enolase (NSE) | at inclusion
  Between group comparison of salivary levels of specific neuronal enolase (NSE) in the 3 groups
Salivary levels of GFAP | at inclusion
  Between group comparison of salivary levels of GFAP in the 3 groups
In vitro fluorescence ratio Dapi / phalloidin | at inclusion
  The fluorescence ratio Dapi / phalloidin in a culture of neurovascular cells in the presence of the serum of the subjects (in vitro) in the 3 groups

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Courtet, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University hospital, Montpellier, France